CLINICAL TRIAL: NCT04434391
Title: Quantitative Fluorescence Polymerase Chain Reaction (QF-PCR) in Group B Strep (GBS) Rectovaginal Colonization Diagnosis During Pregnancy.
Brief Title: QF-PCR In GBS Diagnosis During Pregnancy
Acronym: QFPCRIGDDP
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QF-PCR in GBS screening
Record Dates: First submitted 2013-07-18; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2013-12

CONDITIONS: GBS
Keywords: GBS screening; pregnancy outcome; QF-PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- QF-PCR for GBS screening: QF-PCR for vaginal-rectal samples in pregnant women
  Interventions: Other: QF-PCR for GBS screening

INTERVENTIONS:
Other: QF-PCR for GBS screening — QF-PCR for GBS screening in pregnant women,compared with GBS culture test.

SUMMARY:
Estimate the sensitivity and specificity of Quantitative Fluorescence Polymerase Chain Reaction (QF-PCR) in diagnosing Group B Strep (GBS) rectovaginal colonization during pregnancy, and follow the outcome of the mothers and infants. According to the outcome of this study,the investigator wish to determine that wether QF-PCR is an appropriate screening method for GBS in primary hospitals in China.

DETAILED DESCRIPTION:
This is a study which include 300 pregnant women who will deliver their babies in PUMCH.

1. Obtain vaginal and rectal swab for Group B Strep (GBS) culture and Quantitative Fluorescence Polymerase Chain Reaction (QF-PCR) test between 35-37 weeks.
2. Obtain intrauterine swabs of the woman whose vaginal-rectal GBS test is positive,for both GBS culture and GBS QF-PCR.
3. Obtain rectal and pharynx swabs of the newborns of the woman whose vaginal-rectal GBS test is positive,for both GBS culture and GBS QF-PCR.
4. Blood test for GBS culture and GBS QF-PCR will be carried out to all the babies transferred to neonatal intensive care unit(NICU).
5. For all the samples that GBS culture result was not consistent with QF-PCR, We will do gene sequencing for verification.
6. Pregnant outcome will be followed such as Apgar score,neonatal pneumonia, urinary tract infection, chorioamnionitis, endometritis,sepsis, and bacteremia,It also can cause focal infections such as pneumonia, meningitis, and endocarditis.

Inclusion Criteria:

1.Singleton gestation.Pregnant women between 35-37 weeks gestation. 2.22 years of age or older. 3.Plan to deliver baby in Peking Union Medical College Hospital (PUMCH).

Exclusion Criteria:

1. Preexisting morbidity: Immunocompromised status (HIV +; malignancy; history of organ transplant; chronic steroid therapy; autoimmune disease requiring treatment during pregnancy, and other immunocompromised states); Type 1 diabetes and type 2 diabetes;congenital cardiac disease and cardiac valvular disease requiring antibiotic prophylaxis during procedure/labor; pulmonary disease; renal disease; chronic hepatic disease; inflammatory bowel disease; stomach or duodenal ulcer; bowel resection, gastric bypass, and chronic indwelling venous, bladder, or gastric catheter.
2. Multi-fetal gestation.
3. Chronic (daily) use of broad spectrum antibiotics. 4。Prolonged antibiotic use (> 7 days) in the 4 weeks prior to GBS culture screening.

5.History of infant with GBS sepsis. 6.intrauterine growth retardation(IUGR), Fetal Anomalies-major diagnosed at time of second trimester anatomy ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* 1.Singleton gestation.Pregnant women between 35-37 weeks gestation. 2.22 years of age or older. 3.Plan to deliver baby in PUMCH.

Exclusion Criteria:

* 1.Preexisting morbidity: Immunocompromised status (HIV +; malignancy; history of organ transplant; chronic steroid therapy; autoimmune disease requiring treatment during pregnancy, and other immunocompromised states); Type 1 diabetes and type 2 diabetes;congenital cardiac disease and cardiac valvular disease requiring antibiotic prophylaxis during procedure/labor; pulmonary disease; renal disease; chronic hepatic disease; inflammatory bowel disease; stomach or duodenal ulcer; bowel resection, gastric bypass, and chronic indwelling venous, bladder, or gastric catheter.

  2.Multi-fetal gestation. 3.Chronic (daily) use of broad spectrum antibiotics. 4.Prolonged antibiotic use (> 7 days) in the 4 weeks prior to GBS culture screening.

  5.History of infant with GBS sepsis. 6.IUGR, Fetal Anomalies-major diagnosed at time of second trimester anatomy ultrasound。 7.Anticipated delivery <35 wks for maternal/fetal indication 8.Placenta previa or accreta (with anticipated delivery prior to 35 weeks)

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion Criteria:
  * 1.Singleton gestation.Pregnant women between 35-37 weeks gestation. 2.22 years of age or older. 3.Plan to deliver baby in PUMCH.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with positive results of GBS culture or/and QF-PCR | 3 months
  The percentage will be calculated separately as follows:
  1. Number of positive GBS culture from vaginal/rectal swabs in all participants;
  2. Number of positive GBS QF-PCR from vaginal/rectal swabs in all participants;
  3. Number of positive GBS culture/QF-PCR from intrauterine swabs in women whose vaginal-rectal GBS test is positive;
  4. Number of positive GBS culture from pharynx/rectal swabs in newborns whose mother 's vaginal-rectal GBS test is positive;
  5. Number of positive GBS QF-PCR from pharynx/rectal swabs in newborns whose mother 's vaginal-rectal GBS test is positive;

SECONDARY OUTCOMES:
Number of participants with adverse outcomes of pregnancy | 3 months
  Compare the maternal ante- intra- and postpartum outcomes (urinary tract infections, chorioamnionitis, endometritis, cellulitis, bacteremia, sepsis, and other infectious morbidity) and neonatal outcomes (gestational age at delivery, APGAR scores, bilirubin levels, C-reactive protein, rule out sepsis evaluation, sepsis, pneumonia, meningitis, neonatal ICU admission, and length of hospital stay).

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun MA, MD, Study Director — Peking Union Medical College
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China